CLINICAL TRIAL: NCT06739317
Title: •Stereotactic Body Radiotherapy Combined with Camrelizumab and Apatinib As Conversion Therapy Versus Camrelizumab Combined with Apatinib As First-Line Therapy for Unresectable Hepatocellular Carcinoma: a Prospective, Multicenter, Open-label, Randomized Controlled Clinical Trial.
Brief Title: SBRT Combined with Camrelizumab and Apatinib for Conversion Therapy in Patients with Unresectable Hepatocellular Carcinoma.
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-HCC-II/III-030
Record Dates: First submitted 2024-12-04; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Unresectable Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Radiation: Radiation; Drug: First line therapy; Procedure: operation
- control group (Active Comparator)
  Interventions: Drug: First line therapy

INTERVENTIONS:
Radiation: Radiation — Subjects receive Stereotactic Body Radiotherapy combined with Camrelizumab and Apatinib as conversion therapy.
  Arms: Experimental group
Drug: First line therapy — Subjects receive Camrelizumab intravenously. Subjects receive Apatinib orally.
  Arms: control group
Drug: First line therapy — Subjects receive Camrelizumab intravenously. Subjects receive Apatinib orally.
  Arms: Experimental group
Procedure: operation — If subjects suitable for hepatic resection after conversion therapy, radical surgery and postoperative adjuvant therapy will be performed.
  Arms: Experimental group

SUMMARY:
•This is a randomized, open-label, multi-center, phases 2 and phase 3 trial to evaluate the efficacy and safety of SBRT combined with Camrelizumab and Apatinib as conversion therapy versus Camrelizumab combined with Apatinib as first-Line therapy for unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF).
* Aged 18 years or older.
* Hepatocellular carcinoma confirmed by histology/cytology. Cirrhosis meets the clinical diagnostic criteria for hepatocellular carcinoma of the American Association for the Diagnosis of Liver Diseases (AASLD).
* Barcelona Clinic Liver Cancer stage B or C disease, which was not amenable to radical surgery.
* ECOG Performance Status of 0 or 1.
* Child-Pugh class of A.

Exclusion Criteria:

* Known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and lamellar cell carcinoma; other active malignant tumor except HCC within 5 years or simultaneously.
* Existence of active autoimmune disease or history of autoimmune disease and may relapse.
* Patients with innate or acquired immune deficiency (e.g., HIV infection).
* Known allergies to study drugs or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to approximately 3 years
  The primary endpoint of phase 3 study is OS
The R0 Resection rate of the experimental group | Up to approximately 30 days
  The primary endpoint of phase 2 study is the R0 Resection rate of the experimental group

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 3 years
  The ORR is assessed by the investigators according to RECIST v1.1 and mRECIST, respectively.
Disease control rate (DCR) | Up to approximately 3 years.
  The DCR is assessed by the investigators according to RECIST v1.1 and mRECIST, respectively.
Time to Response (TTR) | Up to approximately 3 years.
  The TTR is assessed by the investigators according to RECIST v1.1 and mRECIST, respectively.
Duration of response (DoR) | Up to approximately 3 years.
  The DoR is assessed by the investigators according to RECIST v1.1 and mRECIST, respectively.
Time to progression (TTP) | Up to approximately 3 years.
  The TTP is assessed by The investigators according to RECIST v1.1 and mRECIST,
Event free survival (EFS) | Up to approximately 3 years.
  The EFS is assessed by the investigators according to RECIST v1.1 and mRECIST, respectively.
Conversion rate | Up to approximately 30 days.
  The conversion rate of the experimental group.
Resection rate | Up to approximately 30 days.
  The resection rate of the experimental group.
R0 resection rate | Up to approximately 30 days.
  The R0 resection rate of the experimental group.
Pathologic complete response (pCR) rate | Up to approximately 30 days.
  The pCR rate of the experimental group.
Major pathological response (MPR) | Up to approximately 30 days.
  The MPR rate of the experimental group.
Safety | Up to approximately 90 days.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No